CLINICAL TRIAL: NCT02384070
Title: Evaluation of Simplified Anti-Thrombotic Therapy for Coronary Fractional Flow Reserve
Brief Title: Simplified Anti-Thrombotic Therapy for FFR
Acronym: SMART-FFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odessa Heart Institute (Other)
Responsible Party: Principal Investigator, Fernando Boccalandro MD, MD FACC FSACI, Odessa Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 20095
Record Dates: First submitted 2015-02-22; First posted 2015-03-10 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Fractional Flow Reserve, Myocardial; Aspirin; Clopidogrel; bivalirudin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Received upstream aspirin plus clopidogrel with no intra-procedural anticoagulation for the FFR calculation with a saline bolus and drip used for placebo anticoagulation during the procedure to blind the operator
  Interventions: Procedure: FFR; Drug: Aspirin; Drug: Clopidogrel
- Group 2 (Active Comparator): Received upstream aspirin and clopidogrel plus intra-procedural anticoagulation with bivalirudin for FFR calculation
  Interventions: Procedure: FFR; Drug: Aspirin; Drug: Clopidogrel; Drug: Bivalirudin
- Group 3 (Experimental): Received only upstream single anti-platelet therapy with aspirin plus intra-procedural anticoagulation for the FFR calculation with bivalirudin
  Interventions: Procedure: FFR; Drug: Aspirin; Drug: Bivalirudin

INTERVENTIONS:
Procedure: FFR — Fractional flow reserve tracings were calculated using a Volcano pressure wire intra-coronary system after ensuring proper calibration of the aortic pressure transducer and the guidewire, using 6 Fr-guide catheters. Before crossing the stenosis, baseline pressure was measured by the guide catheter and the pressure guidewire were equalized according to the manufacturer's specifications. After advancing the pressure sensor across the stenosis, coronary hyperemia was induced using intravenous adenosine (140μg/kg/min until a steady state was reached for at least 3 minutes). Fractional flow reserve was considered positive if it was less than 0.80.
  Other Names: Fractional Flow Reserve
Drug: Aspirin — All patients received a chewable aspirin of 325 mg at least 6 hours before the procedure
Drug: Clopidogrel — All patient receiving clopidogrel, were loaded with 600 mg at least 6 hours before the procedure
  Arms: Group 1; Group 2
Drug: Bivalirudin — Dosed based on the weight at 0.75 mg/kg I.V. bolus dose followed by a 1.75 mg/kg/hr I.V. infusion for the duration of the procedure
  Arms: Group 2; Group 3

SUMMARY:
Despite the routine use of procedural anti-coagulation and anti-platelet therapy for FFR calculation, no study has evaluated the optimal anti-thrombotic regimen in patients undergoing FFR. Therefore, the aim of the Evaluation of Simplified Anti-Thrombotic Therapy for Coronary Fractional Flow Reserve (SMART-FFR) study was to evaluate the safety of using a simplified anti-thrombotic regimen with only upstream dual anti-platelet therapy (DAT) with aspirin and clopidogrel, compared with anticoagulation plus single- or- DAT therapy in patients with intermediate coronary artery stenosis undergoing FFR calculation during elective coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* All patient regardless of sex, or age were eligible for the study if they were scheduled for an elective coronary angiography using a femoral approach, and were agreeable to participate in the study after signing informed consent, and had a coronary stenosis in any major native epicardial coronary artery between 50-70% determined by quantitative angiography that was an adequate target for FFR at the discretion of the operator.

Exclusion Criteria:

* Exclusion criteria included patients requiring mandatory DAT, patient undergoing radial access due to concomitant anticoagulation, patients with contra-indications or intolerant to DAT, patients with severe left ventricular hypertrophy defined as a wall thickness greater than 14 mm by echocardiography in the septal or lateral wall, patients with hypertrophic cardiomyopathy, left ventricular function less than 30%, severe aortic valvular stenosis defined as an aortic valve area of less than 1 cm2, presenting with an acute coronary syndrome in the past two weeks, hemodynamic instability, cardiogenic shock, reported allergy to clopidogrel, aspirin or bivalirudin, planned to be anticoagulated during or previous to the time of the coronary angiography, using Prasugrel or Ticagrelor, patients with coronary arteries unsuitable for FFR calculation due to severe tortuousity and/or calcification, lesions supplied by a bypass conduit, any mental condition rendering the subject incapable to understand the nature, scope, and possible consequences of the study such that the patient is unable to give appropriate informed consent or refusal or inability to sign an informed consent .

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Upstream Aspirin + Clopidrogel: Received upstream aspirin plus clopidogrel with no intra-procedural anticoagulation for the FFR calculation with a saline bolus and drip used for placebo anticoagulation during the procedure to blind the operator
- Group 2: Upstream Aspirin and Clopidrogel Plus Bivalirudin: Received upstream aspirin and clopidogrel plus intra-procedural anticoagulation with bivalirudin for FFR calculation
- Group 3: Upstream Aspirin Plus Bivalirudin: Received only upstream single anti-platelet therapy with aspirin plus intra-procedural anticoagulation for the FFR calculation with bivalirudin
Period: Overall Study
Arm/Group | Group 1: Upstream Aspirin + Clopidrogel | Group 2: Upstream Aspirin and Clopidrogel Plus Bivalirudin | Group 3: Upstream Aspirin Plus Bivalirudin
Started | 100 | 100 | 100
Completed | 100 | 100 | 100
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Upstream Aspirin + Clopidrogel: Aspirin: All patients received a chewable aspirin of 325 mg at least 6 hours before the procedure
  Clopidogrel: All patient receiving clopidogrel, were loaded with 600 mg at least 6 hours before the procedure
- Group 2: Upstream Aspirin and Clopidrogel Plus Bivalirudin: Aspirin: All patients received a chewable aspirin of 325 mg at least 6 hours before the procedure
  Clopidogrel: All patient receiving clopidogrel, were loaded with 600 mg at least 6 hours before the procedure
  Bivalirudin: Dosed based on the weight at 0.75 mg/kg I.V. bolus dose followed by a 1.75 mg/kg/hr I.V. infusion for the duration of the procedure
- Group 3: Upstream Aspirin Plus Bivalirudin: Aspirin: All patients received a chewable aspirin of 325 mg at least 6 hours before the procedure
  Bivalirudin: Dosed based on the weight at 0.75 mg/kg I.V. bolus dose followed by a 1.75 mg/kg/hr I.V. infusion for the duration of the procedure
- Total: Total of all reporting groups
Arm/Group | Group 1: Upstream Aspirin + Clopidrogel | Group 2: Upstream Aspirin and Clopidrogel Plus Bivalirudin | Group 3: Upstream Aspirin Plus Bivalirudin | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (9) | 65 (10) | 63 (8) | 64 (3)
Gender [Count of Participants; unit: Participants]
  Female | 38 | 39 | 35 | 112
  Male | 62 | 61 | 65 | 188
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 100 | 300

OUTCOME MEASURES:

1. Primary Outcome: Thrombotic Complications
Time Frame: Hospital Stay and after 30 days post PCI
Measure: Number; unit: Number of Patients
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 100 | 100 | 100
Number of Patients | 0 | 0 | 0
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Superiority or Other; p = 1, ANOVA — Analysis of the variance was used and Chi-square test for categorical variables. A sample size was calculated for a 95% confidence level and a power of 80%, assuming a 10% difference between groups
Statistical Analysis 2: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Superiority or Other; p = 1, ANOVA — The prior threshold for statistical significance was P < 0.05

2. Secondary Outcome: TIMI (Thrombolysis in Myocardial Infarction) Major and Minor Bleeding Scores
Description: 1. Major: Intracranial bleeding, Clinically overt signs of hemorrhage associated with a drop in hemoglobin of ≥5 g/dL or a ≥15% absolute decrease in haematocrit or Fatal bleeding.
  2. Minor: Clinically overt (including imaging), resulting in hemoglobin drop of 3 to <5 g/dL or ≥10% decrease in haematocrit. No observed blood loss: ≥4 g/dL decrease in the haemoglobin concentration or ≥12% decrease in haematocrit Any overt sign of hemorrhage that meets one of the following criteria and does not meet criteria for a major or minor bleeding event, as defined above Requiring intervention
Time Frame: Hospital Stay and after 30 days post PCI
Measure: Number; unit: Patients
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 100 | 100 | 100
Patients | 1 | 3 | 1

3. Secondary Outcome: Sub-clinical Ischemic Events Measured by Troponin Levels Post-procedure
Time Frame: 48 hours post procedure
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 100 | 100 | 100
participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No